CLINICAL TRIAL: NCT03169400
Title: Molecular and Cellular Mechanism of Vascular Ageing in Chronic Kidney Disease: Role of Theranova Dialyzer on Mineral Metabolism Disorder, Oxidative Stress, and Vascular Calcification
Brief Title: Theranova Dialyzer and Chronic Kidney Disease - Mineral Bone Disorder (CKD-MBD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Mario Cozzolino, Professor of Nephrology, MD, PhD, FERA, FASN, University of Milan
Other Study IDs: BXT-MI1
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: End Stage Renal Failure on Dialysis; Vascular Calcification; Oxidative Stress
Keywords: vascular calcification; haemodialysis; dialysis membrane
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Theranova treated: We will collect pool of human sera from HD patients treated with regular bicarbonate dialysis membrane (baseline). Then, patients will be treated for 3 months with Theranove dialyzer, and sera will be collected at 1, 2, and 3 months. We will create a serum pool.
  Interventions: Device: Theranova dialyzer
- Standard treated: We will collect pool of human sera from HD patients treated with regular bicarbonate dialysis membrane (baseline). Then, patients will be treated for 3 months with Theranove dialyzer, and sera will be collected at 1, 2, and 3 months. We will create a serum pool.

INTERVENTIONS:
Device: Theranova dialyzer — Hemoadialysis
  Other Names: Theranova
  Groups: Theranova treated

SUMMARY:
The project will be structured in 3 main parts:

1. Effect of sera of ESRD patients on HD using Theranova dialyzer on high-Pi induced vascular calcification in an in vitro model of rat VSMCs.
2. Effect of sera of ESRD patients on HD using Theranova dialyzer on oxidative stress pathways in an in vitro model of rat VSMCs vascular calcification.
3. Study of RNA sequencing, transcriptome analysis gene expression of time course high-P challenged VSMCs studying the effect of sera of ESRD patients on HD using Theranova dialyzer

DETAILED DESCRIPTION:
Ageing is a potent, independent risk factor for cardiovascular (CV) disease and the calcification of the vascular smooth muscle cell (VSMC) layer of the vessel media, typical of Monckenberg syndrome, is a hallmark of vascular ageing. Young patients with chronic kidney disease (CKD) exhibit an extremely high CV mortality, equivalent to that seen in octogenarians in the general population. Even children on dialysis develop accelerated medial vascular calcification (VC) and arterial stiffening, leading to the suggestion that patients with CKD exhibit a 'premature ageing' phenotype. It is now well documented that uraemic toxins, particularly those associated with dysregulated mineral metabolism, can drive VSMC damage and phenotypic changes that promote VC, and epidemiological data suggest that some of these same risk factors associate with CV mortality in the aged general population.

VC is common in CKD and associated with increased morbidity and mortality. Its mechanism is multifactorial and incompletely understood. CKD patients are at risk for VC because of multiple risk factors that induce VSMCs to change into a osteoblast-like cell such as high total body burden of calcium (Ca) and phosphorus (P) due to abnormal bone metabolism, low levels of circulating and locally produced inhibitors, impaired renal excretion, and current therapies. Together these factors increase risk and complicate the management of VC. Cells with unexpected osteoblastic potential may abnormally lay down some forms of VC, especially in the arterial wall of blood vessels. The pathogenesis of VC is likely a hybrid process of tightly regulated normal bone modeling and the purely physicochemical deposition of mineral.

The interest in VC in CKD patients has several reasons. First, it is now clear that in the general population the calcification of both intimal atherosclerotic lesions and the medial vessel layer are associated with CV morbidity and mortality. Similar, some data also exists for stage 5 CKD. Second, there is now better evidence that VSMCs can become osteoblast-like and lay down and mineralize collagen and noncollagenous proteins in arteries. Third, over 20 null mutations in mice have VC confirming that key proteins regulate or prevent VC. Fourth, there is increasing recognition of a link between CKD and bone and VC in the general population. Lastly, we now know some of our well-intended interventions to treat renal osteodystrophy accelerate arterial calcification.

CKD patients have an increased CV risk factor due to the impaired renal function induced by the pathology. More than 90% of CKD patients die for CV events with a main role of VC. One of the VC inducer is HD per se. Since the choice of dialyzer may play a role on prevalence of CV complication in CKD, the aim of this project will be to elucidate the effect of Theranova dialyzer on delay VC progression.

The project will be structured in 3 main parts:

1. Effect of sera of ESRD patients on HD using Theranova dialyzer on high-Pi induced vascular calcification in an in vitro model of rat VSMCs.
2. Effect of sera of ESRD patients on HD using Theranova dialyzer on oxidative stress pathways in an in vitro model of rat VSMCs vascular calcification.
3. Study of RNA sequencing, transcriptome analysis gene expression of time course high-P challenged VSMCs studying the effect of sera of ESRD patients on HD using Theranova dialyzer Primary Endpoint: Effect of sera of ESRD patients on HD using Theranova dialyzer on high-Pi induced vascular calcification in an in vitro model of rat VSMCs.

Secondary Endpoints: Effect of sera of ESRD patients on HD using Theranova dialyzer on oxidative stress pathways in an in vitro model of rat VSMCs vascular calcification.

Study of RNA sequencing, transcriptome analysis gene expression of time course high-P challenged VSMCs studying the effect of sera of ESRD patients on HD using Theranova dialyzer

ELIGIBILITY:
Key Inclusion Criteria: ESRD on HD

Key Exclusion Criteria: cachexia; cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients
  Number of study or comparison groups: cross-over study; from HD patients treated with regular bicarbonate dialysis membrane (baseline). Then, patients will be treated for 3 months with Theranove dialyzer, and sera will be collected at 1, 2, and 3 months. We will create a serum pool.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of sera of ESRD patients on HD using Theranova dialyzer on high-Pi induced vascular calcification in an in vitro model of rat VSMCs. | 12 months
  Quantification of calcium into the cells

SECONDARY OUTCOMES:
Effect of sera of ESRD patients on HD using Theranova dialyzer on oxidative stress pathways in an in vitro model of rat VSMCs vascular calcification. | 12 months
  Oxidative stress into the cells

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No